CLINICAL TRIAL: NCT03800745
Title: Reduction of Postoperative Gastrointestinal Dysmotility Following Total Laparoscopic Hysterectomy: a Randomized Control Trial.
Brief Title: Reduction of Postoperative Gastrointestinal Dysmotility Following Total Laparoscopic Hysterectomy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Michael Sprague MD (Unknown); Pamela Frazzini-Padilla MD (Unknown); Katherine Smith MD (Unknown); Jennifer Afton Cooper MD (Unknown)
Responsible Party: Principal Investigator, Mehandru, Natasha, Sub-Investigator; Study Coordinator, The Cleveland Clinic
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FLA 18-069
Record Dates: First submitted 2019-01-08; First posted 2019-01-11 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Postoperative Passage of Flatus; Postoperative Bowel Movement
MeSH Terms: interventions — Dioctyl Sulfosuccinic Acid; polyethylene glycol 3350

STUDY DESIGN:
Intervention Model Description: randomized control trial
Masking Description: Participants are randomized to their arm on the day of surgery. A manila envelope with the arm written on a paper inside the envelope is opened in the post-anesthesia care unit (PACU) following surgery. A computerized random number generator was used to assign arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- No Medication (No Intervention): No intervention is assigned in Arm A.
- Colace (Experimental): This is Arm B. Docusate sodium(Colace) is prescribed as100mg twice daily orally. Patients will be instructed to begin taking this the evening of surgery through postoperative day five.
  Interventions: Drug: Colace 100Mg Capsule
- Miralax (Experimental): This is Arm C. Miralax 17 grams oral powder pack daily is prescribed to be taken with breakfast. Patients will be instructed to begin taking this the morning after surgery through postoperative day five.
  Interventions: Drug: Miralax

INTERVENTIONS:
Drug: Colace 100Mg Capsule — Prescribed to Arm B
  Arms: Colace
Drug: Miralax — Prescribed to Arm C
  Arms: Miralax

SUMMARY:
Return of bowel function is an integral component of postoperative recovery following minimally invasive gynecologic surgery. To date, there is no standardized regimen to optimize bowel motility postoperatively. Clinical practices vary in the medications prescribed to facilitate this process, as well as what is considered the norm for return of flatus and time to first bowel movement.

This study is a randomized control trial. The primary outcome of the study is to assess the effect of a standardized postoperative bowel care regimen on return of bowel function by assessing the time to first bowel movement; a secondary outcome is to assess the effect of such a regimen on time to first flatus. The hypothesis is that the prescription of a laxative, rather than a stool softener or no agent, will expedite the time to first bowel movement and first flatus. Other secondary outcomes and endpoints are assessing narcotic use measured in total oral morphine equivalents in the first five days postoperatively, as well as the constipation score and the PAC-SYM questionnaire.

DETAILED DESCRIPTION:
Patients undergoing minimally invasive hysterectomy at Cleveland Clinic Florida Department of Minimally Invasive Gynecologic Surgery will be recruited at their preoperative visit or over the phone. Inclusion criteria will be patients aged 18-85 undergoing minimally invasive gynecologic surgery in the form of total laparoscopic hysterectomy. Exclusion criteria are an underlying gynecologic malignancy, pre-existing gastrointestinal disorders, history of bowel resection, insulin-dependent diabetes or gastroparesis, known gastric dysmotility, chronic use of pain medications, or anticipated bowel surgery. Subjects that routinely take laxatives will be included in a sub-analysis. Randomization will occur in the immediate postoperative period. Enrolled subjects will be randomized using a computer generator. A total sample size of 72 subjects, with 24 subjects in each arm, is needed to attain a significance level of 95% at a power of 80% to demonstrate a reduction of 24 hours or more to first postoperative bowel movement. Accounting for a 10% attrition rate, we will aim to recruit 81 patients total with 27 subjects in each arm. The control group, arm A, will be not be prescribed any postoperative bowel care regimen. The first study group, arm B, will be prescribed docusate sodium(Colace) 100mg twice daily orally, and will be instructed to begin taking this the evening of surgery through postoperative day five. One dose will be taken with breakfast every morning, and the second dose will be taken with dinner every evening. The second study group, arm C, will be prescribed Miralax 17 grams oral powder pack daily with breakfast, and will be instructed to begin taking this the morning after surgery through postoperative day five. Prescriptions will be given at the time of randomization immediately postoperatively and prior to discharge home. At Cleveland Clinic Florida, a majority of patients are discharged the day of surgery.

In addition, the presence of preoperative constipation will be assessed prior to surgery based on the Rome IV criteria along with baseline stool consistency as per the Bristol Stool Chart. Postoperatively, patients will be asked to record the time of first flatus and time first bowel movement. Each subject will complete the Patient Assessment of Constipation Symptoms (PAC-SYM) validated questionnaire on postoperative day 5, and a constipation score will also be calculated. Compliance with postoperative medications will also be assessed as defined by the number of medications taken as prescribed. Patients will record medications taken each day in a medication diary.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-85 undergoing minimally invasive gynecologic surgery in the form of total laparoscopic hysterectomy.

Exclusion Criteria:

* an underlying gynecologic malignancy, pre-existing gastrointestinal disorders, history of bowel resection, insulin-dependent diabetes or gastroparesis, known gastric dysmotility, chronic use of pain medications, or anticipated bowel surgery

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Time to First Bowel Movement | Patients will be followed for the first 5 days after surgery.
  The primary outcome of the study is to assess the effect of a standardized postoperative bowel care regimen on return of bowel function by assessing the date and time of first BM after surgery.

SECONDARY OUTCOMES:
Time to First Flatus | Patients will be followed for the first 5 days after surgery.
  Secondary outcomes include the time to first flatus. This will be calculated as the difference between the date and end time of the subject's surgery and the date and time of first BM after surgery.
Narcotic Use | Patients will be followed for the first 5 days after surgery.
  Postoperative narcotic use in oral morphine equivalents in the first five days postoperatively will be measured.
PAC-SYM Questionnaire | Patients will be followed for the first 5 days after surgery.
  To assess for opioid-induced constipation. Postoperatively, the Patient Assessment of Constipation-Symptom Questionnaire will be administered on postoperative day 5 to assess 12 different symptoms regarding bowel function.The 12-item questionnaire is divided into three symptom subscales: abdominal (four items); rectal (three items); and stool (five items). Items are scored on 5-point Likert scales, with scores ranging from 0 to 4 (0 = 'symptom absent', 1 = 'mild', 2 = 'moderate', 3 = 'severe' and 4 = 'very severe'). A mean total score in the range of 0-4 is generated by dividing the total score by the number of questions completed; the lower the total score, the lower the symptom burden. Historically, a reduction in total score of 1 point or more has been used as the cut-off to define a positive response to treatment, 2 implying that this is a meaningful improvement.
Constipation Score | The first 5 days after surgery.
  A postoperative constipation score is calculated based on preoperative stool frequency, postoperative days to first BM, stool consistency, percentage of straining, and sensation of incomplete evacuation. Constipation scores are calculated basedon: days to first BM (2 points if >4 days, 0 points if 1-3 days); stool consistency (1 point if types 1 or 2, 0 points for types 3-7); strain rating (0.5 points if for ≥5 on ≥25% of the BMs; 0 points for ≤4 on 0-25%); 0.5 point for rating of mild, moderate, or severe for sense of incomplete evacuation to the question: "Have you experienced incomplete bowel movement, like you did not finish?" with 0 point for rating of none). The Straining Scale is a single-item questionnaire assessing straining on a 5 point Likert scale ranging from 1 to 5 in the following order: no straining, mild, moderate, severe, or very severe straining. A constipation score of 2 or more is consistent with constipation based on the Rome III criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No